CLINICAL TRIAL: NCT00350389
Title: Randomised Controlled Falls Prevention Trial of Plain Distance Glasses in Elderly Multifocal Wearers.
Brief Title: VISIBLE Study (Visual Intervention Strategy Incorporating Bifocal & Long-distance Eyewear)
Acronym: VISIBLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: South Eastern Area Health Service (Other); Northern Sydney and Central Coast Area Health Service (Other)
Responsible Party: Principal Investigator, Stephen Lord, Senior Principal Research Fellow, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 350855
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Falls
Keywords: Falls, Older persons
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Provision of single lens glasses, glasses aids, counselling, updated multifocal glasses if required
  Interventions: Behavioral: Outdoor use of plain distance glasses with counselling
- 2 (No Intervention): Usual care, updated multifocal glasses if required

INTERVENTIONS:
Behavioral: Outdoor use of plain distance glasses with counselling — Provision of single lens glasses, glasses aids, counselling, updated multifocal glasses if required
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether the provision of supplementary plain distance glasses for outdoor use to older users multifocal glasses will reduce falls rates over a 12 month period.

DETAILED DESCRIPTION:
Background: Bi-, tri- and multi- focal ('multifocal') glasses have been associated with increased rates of falls in older people (Lord et al 2002).

Study Aim: To determine whether the provision of supplementary plain distance glasses for outdoor use to older users multifocal glasses will reduce falls rates over a 12 month period.

Study Design: A randomised controlled assessor-blinded trial with two parallel groups in 580 participants. Study inclusion criteria are: outdoor use of multifocal glasses 3 or more times per week, community-dwelling persons aged 65+ years with a recent fall OR persons aged 80+ years regardless of falls history, Folstein Mini Mental score of 24+, and adequate visual contrast sensitivity (Melbourne Edge Test score of 16+dB). All participants will receive an optometry assessment and updated multifocal glasses (if required) at baseline. Intervention group subjects will receive a pair of plain distance glasses and counselling for their use in predominantly outdoor situations. Control group participants will use their multifocal glasses in their usual manner. Falls rates and compliance with the intervention will be recorded on monthly falls diaries returned by the participants.

ELIGIBILITY:
Inclusion Criteria:

* outdoor use of multifocal glasses 3 or more times per week
* community-dwelling persons aged 65+ years with a recent fall OR persons aged 80+ years regardless of falls history
* Folstein Mini Mental score of 24+
* adequate visual contrast sensitivity (Melbourne Edge Test score of 16+dB)

Exclusion Criteria:

* nursing home residents

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 606 (Actual)
Dates: Start 2005-06; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Falls rates, Falls diaries | 12 months

SECONDARY OUTCOMES:
Quality of life, SF-36 | 12 months
Instrumental Activities of Daily Living, Adelaide Activities Profile | 12 months
Modified Falls Efficacy Scale | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Lord, PhD, Principal Investigator — University of New South Wales
Locations (1):
- Prince of Wales Medical Research Institute, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Lord SR, Dayhew J, Howland A. Multifocal glasses impair edge-contrast sensitivity and depth perception and increase the risk of falls in older people. J Am Geriatr Soc. 2002 Nov;50(11):1760-6. doi: 10.1046/j.1532-5415.2002.50502.x. PMID 12410892
- [Derived] Clemson L, Stark S, Pighills AC, Fairhall NJ, Lamb SE, Ali J, Sherrington C. Environmental interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2023 Mar 10;3(3):CD013258. doi: 10.1002/14651858.CD013258.pub2. PMID 36893804
- [Derived] Haran MJ, Cameron ID, Ivers RQ, Simpson JM, Lee BB, Tanzer M, Porwal M, Kwan MM, Severino C, Lord SR. Effect on falls of providing single lens distance vision glasses to multifocal glasses wearers: VISIBLE randomised controlled trial. BMJ. 2010 May 25;340:c2265. doi: 10.1136/bmj.c2265. PMID 20501583
- [Derived] Haran MJ, Lord SR, Cameron ID, Ivers RQ, Simpson JM, Lee BB, Porwal M, Kwan MM, Severino C. Preventing falls in older multifocal glasses wearers by providing single-lens distance glasses: the protocol for the VISIBLE randomised controlled trial. BMC Geriatr. 2009 Mar 26;9:10. doi: 10.1186/1471-2318-9-10. PMID 19321012